CLINICAL TRIAL: NCT01217762
Title: A Pilot Study to Evaluate the Safety and Tolerability of the IRay Stereotactic Radiosurgery System in Subjects With Exudative Choroidal Neovascularization (CNV) Secondary to Age-Related Macular Degeneration (AMD)
Brief Title: Safety & Tolerability of the IRay System in Subjects With Exudative Choroidal Neovascularization (CNV) Secondary to Age-Related Macular Degeneration (AMD)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oraya Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLH001
Record Dates: First submitted 2010-10-05; First posted 2010-10-08 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2012-01

CONDITIONS: Age-Related Macular Degeneration; Wet Age-Related Macular Degeneration; Macular Degeneration; Eye Diseases; Retinal Diseases
Keywords: Oraya; Oraya Therapeutics, Inc.; low voltage stereotactic radiosurgery; radiosurgery; radiotherapy; IRay; AMD; Macular Degeneration; Wet AMD; xray; radiation; x ray; external beam radiation; Ranibizumab; Lucentis
MeSH Terms: conditions — Macular Degeneration; Eye Diseases; Retinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 11 Gy IRay (Experimental): Day 0 Lucentis followed by 11 Gy IRay, Lucentis at Month 1 and Lucentis PRN (N = 2)
  Interventions: Device: IRay
- 16 Gy IRay (Experimental): Day 0 Lucentis followed by 16 Gy IRay, Lucentis at Month 1 and Lucentis PRN (N = 27)
  Interventions: Device: IRay
- 16 Gy IRay - Radiation First (Experimental): 16 Gy IRay and Lucentis PRN (N = 13)
  Interventions: Device: IRay
- 24 Gy IRay (Experimental): Day 0 Lucentis followed by 24 Gy IRay, Lucentis at Month 1 and Lucentis PRN (N = 19)
  Interventions: Device: IRay

INTERVENTIONS:
Device: IRay — Low voltage stereotactic radiotherapy system

SUMMARY:
The purpose of this study is to evaluate the safety and clinical feasibility of the IRay System for the treatment of wet age-related macular degeneration (AMD).

DETAILED DESCRIPTION:
The primary objective is to evaluate the safety and clinical feasibility of stereotactic radiotherapy with the Oraya IRay system for the treatment of choroidal neovascularization (CNV) associated with age-related macular degeneration (AMD), as measured by incidence and severity of ocular radiation related serious adverse events (SAE) and adverse events (AE) in subjects treated with an 11, 16 or 24 Gray (Gy) macular dose through the 60-month follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be age 50 or older
* Women must be post-menopausal ≥1 year or surgically sterilized
* Subjects must have choroidal neovascularization lesion size of ≤11 total disc areas (28.26mm), and a greatest linear dimension of ≤6 mm
* Subjects must have Early Treatment Diabetic Retinopathy Study (ETDRS) best corrected visual acuity of 69 to 24 letters (20/40 to 20/320 Snellen Equivalent) in the study eye
* Subretinal hemorrhage (if any) must not comprise more than 50% of total lesion size, and may not involve the subfoveal space

Exclusion Criteria:

* Subjects with prior or concurrent therapies including submacular surgery, thermal laser photocoagulation (with or without photographic evidence), photodynamic therapy and transpupillary thermotherapy (TTT)
* Subjects with concomitant disease in the study eye, including uveitis, diabetic retinopathy,presence of RPE tears or rips, acute ocular or periocular infection
* Subjects with advanced glaucoma (>0.8 cup to disk ratio) or intraocular pressure ≥30 mmHg in the study eye
* Previous glaucoma filtering surgery in the study eye
* Refractive error in the study eye demonstrating more than -8 diopters of myopia (or globe axial length ≥26 mm). For subjects who have undergone prior refractive or cataract surgery in the study eye, the preoperative refractive error cannot exceed -8 diopters of myopia
* Subjects with any retinal vasculopathies, including diabetic retinopathy, retinal vein occlusions, etc. in the study eye

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2008-07; Primary Completion 2010-10 (Actual); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of ocular radiation-related adverse events | Month 12

SECONDARY OUTCOMES:
Incidence of ocular adverse events | Through month 60
Percentage of subjects who lose at least 15 Early Treatment Diabetic Retinopathy Study (ETDRS) letters in best corrected visual acuity (BCVA) | Month 12
Percentage of subjects gaining ≥ 15 ETDRS letters | Month 12
Percentage of subjects gaining ≥ 0 ETDRS letters | Month 12
Mean change in ETDRS visual acuity | Month 12
Mean time to anti-VEGF retreatment following 2nd mandatory injection (excluding radiation-first subjects) | Month 12
Mean total number of ranibizumab injections | Through month 12 and 24
Change in choroidal neovascularization (CNV) size by fluorescein angiography (FA) | Month 12
Change in total lesion size by fluorescein angiography (FA) | Month 12
Change in central retinal lesion thickness by optical coherence tomography (OCT) | Month 12
Change in central subfield thickness by optical coherence tomography (OCT) | Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Denis O'Shaughnessy, Ph.D., Study Director — Oraya Therapeutics, Inc.
Locations (1):
- Asociación Para Evitar la Ceguera en México, I.A.P., Mexico City, Delegación Coyoacán, Mexico

REFERENCES:
- [Derived] Moshfeghi AA, Morales-Canton V, Quiroz-Mercado H, Velez-Montoya R, Zavala-Ayala A, Shusterman EM, Kaiser PK, Sanislo SR, Gertner M, Moshfeghi DM. 16 Gy low-voltage x-ray irradiation followed by as needed ranibizumab therapy for age-related macular degeneration: 12 month outcomes of a 'radiation-first' strategy. Br J Ophthalmol. 2012 Oct;96(10):1320-4. doi: 10.1136/bjophthalmol-2011-301222. Epub 2012 Aug 15. PMID 22895887